CLINICAL TRIAL: NCT05373394
Title: Evaluation of Cognitive and Motor Neurological Disorders in the Short and Long Term After Surgery for the Removal of a Diffuse Low-grade Glioma of the Supplementary Motor Area
Acronym: POG-C
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR220033
Record Dates: First submitted 2022-05-02; First posted 2022-05-13 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Cognitive Disorders; Motor Disorders; Low-grade Glioma
Keywords: glioma; supplementary motor area; neurological disorders
MeSH Terms: conditions — Cognitive Dysfunction; Motor Disorders; Glioma; Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: patients with a history of surgical removal of diffuse low grade glioma located in the supplementary motor area
  Interventions: Other: Test battery
- Control: patients with a history of surgical removal of diffuse low-grade glioma located in another brain area
  Interventions: Other: Test battery

INTERVENTIONS:
Other: Test battery — motor and neuropsychological test battery

SUMMARY:
Background : The supplementary motor area is the most common/preferential brain location of LGG. This area plays an important role in many motor and cognitive functions such as motor initiation, bimanual coordination and executive functions. Many studies describe the supplementary motor area syndrome resulting from lesions in this area. News managements for LGGs consisting in intraoperative mapping in awake patients reduce significantly neurological disorders and increase also the overall survival . However, the literature does not provide data concerning motor and cognitive functions in a long term and their consequences in the quality of life of patients.

Objective : The aim of our research project is to identify whether there are some motor or neurocognitive deficit in the short and the long term in a population of patients who have medical story of LGG resection in the supplementary motor area.

DETAILED DESCRIPTION:
Patients and Methods : 20 patients who have medical story of LGG in the supplementary motor area and 20 patients who have medical story of LGG resection in other locations are recruited. Firstly, patients have to complete a self-assessment questionnaire about their quality of life, sent by regular mail or e-mail. Then, patients are admitted on the same day as their follow up visit and underwent motor and neurocognitive screening tests ( "Bilan des 400 points", Tests of Attentional Performances) for an hour. The investigators will analyse data and compare between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have a history of low-grade diffuse glioma resection
* Visiting the University Hospital for a follow-up neurosurgical consultation
* Underwent awake surgery

Exclusion Criteria:

* Presence of cognitive disorders that do not allow the proposed test battery to be performed
* Under guardianship or curatorship
* Opposition to the participation to the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with low-grade diffuse glioma resection visiting the university hospital for a follow-up neurosurgical consultation
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
motor tests in the case group - 400 point assessment | inclusion visit
  analysis of the scores obtained at the tests 4 tests :
  * Hand mobility
  * Grip strength
  * Single-handed grasp and movement of objects
  * Two-handed grasp and movement of objects Minimum value = 0 Maximum value = 100 100/100 means that the various tests regain good motor skills and hand grasp
neuropsychological tests in the case group | inclusion visit
  analysis of the scores obtained Phase alert system
  * Reaction time (RT) and standard deviation (SD) measurement with horn
  * Measurement of reaction times (RT) and standard deviation(SD) without horn
  * Measurement of the phase alert index
  Flexibility
  * Measurement of reaction times (RT) and standard deviation (SD) with hand change
  * Measurement of reaction times (RT) and standard deviation (SD) without hand change
  * Overall performance index
  * Speed accuracy trade off index
  * Number of wrong answers
  Incompatibility
  * Measurement of reaction times (RT) and standard deviation (SD) in compatible condition
  * Measurement of reaction times (RT) and standard deviation (SD) in incompatible condition
  * F (visual field)
  * F (hand)
  * F (incompatibility: fields * hand)
  * Number of false responses
  RT min : 0 SD min : 0 No maximum value: calculation against standard values

SECONDARY OUTCOMES:
motor tests in the control group - 400 point assessment | inclusion visit
  analysis of the scores obtained at the tests 4 tests :
  * Hand mobility
  * Grip strength
  * Single-handed grasp and movement of objects
  * Two-handed grasp and movement of objects Minimum value = 0 Maximum value = 100 100/100 means that the various tests regain good motor skills and hand grasp
neuropsychological tests in the control group | inclusion visit
  analysis of the scores obtained Phase alert system
  * Reaction time (RT) and standard deviation (SD) measurement with horn
  * Measurement of reaction times (RT) and standard deviation(SD) without horn
  * Measurement of the phase alert index
  Flexibility
  * Measurement of reaction times (RT) and standard deviation (SD) with hand change
  * Measurement of reaction times (RT) and standard deviation (SD) without hand change
  * Overall performance index
  * Speed accuracy trade off index
  * Number of wrong answers
  Incompatibility
  * Measurement of reaction times (RT) and standard deviation (SD) in compatible condition
  * Measurement of reaction times (RT) and standard deviation (SD) in incompatible condition
  * F (visual field)
  * F (hand)
  * F (incompatibility: fields * hand)
  * Number of false responses
  RT min : 0 SD min : 0 No maximum value: calculation against standard values
Brain MRI | inclusion visit
  Analysis of the location of diffuse low-grade gliomas
Brain MRI | inclusion visit
  Analysis of the lesion volume of diffuse low-grade gliomas
quality of life self-questionnaire carried out at home : sickness Impact Profile | inclusion visit
  analysis of the results obtained 136 questions with responses True or False Minimum value = 0 Maximum value = 136 136/136 means that the quality of life is very negatively affected
fatigue self-questionnaire carried out at home : fatigue Impact Scale (FIS) | inclusion visit
  analysis of the results obtained 40 questions with responses
  * It is quite true
  * It is rather true
  * It is neither true nor false
  * It is rather false
  * It is completely false

CONTACTS AND LOCATIONS:
Overall Officials: Ilyess ZEMMOURA, Principal Investigator — University Hospital, Tours
Locations (1):
- University hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided